CLINICAL TRIAL: NCT05245149
Title: Prospective Observational Study of Image Quality and Radiation Dose Associated With Cardiac Scans in Modern CT Scanners
Brief Title: Image Quality and Radiation Dose Associated With Cardiac Scans in Modern CT Scanners
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Augsburg (Other)
Responsible Party: Sponsor
Other Study IDs: 21-0383
Record Dates: First submitted 2021-07-15; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2021-07

CONDITIONS: Coronary Artery Disease
Keywords: Spectral CT; Multi-Energy CT; Photon Counting Detector CT; PCD-CT
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective Cohort: Patients with a clinical indication for coronary CT angiography will undergo this scan on a photon counting detector CT (PCD-CT).
  Interventions: Diagnostic Test: Cardiac CTA on a photon-counting detector CT (PCD-CT)
- Retrospective Cohort: For comparison, a matched retrospective cohort will be created of patients who had undergone coronary CT angiography on prior CT scanner generations (with energy-integrating detector CT, EID-CT)
  Interventions: Diagnostic Test: Cardiac CTA on a regular CT with Energy-Integrating Detector (EID-CT)

INTERVENTIONS:
Diagnostic Test: Cardiac CTA on a photon-counting detector CT (PCD-CT) — Cardiac CTA will be performed on a dual-source photon-counting CT
  Groups: Prospective Cohort
Diagnostic Test: Cardiac CTA on a regular CT with Energy-Integrating Detector (EID-CT) — Cardiac CTA was performed on a dual-source CT with regular energy-integrating detector (EID-CT)
  Groups: Retrospective Cohort

SUMMARY:
The main objective of this study is to evaluate the dose efficiency of coronary CT angiography (CTA) using a photon counting detector CT (PCD-CT) with the dose efficiency of coronary CT angiography of prior CT generations. 100 patients with a clinical indication for coronary CT angiography will be prospectively enrolled and undergo coronary CTA on a PCD-CT. For comparison, a matched retrospective cohort of 100 patients will be created who had undergone on a prior scanner generation (retrospective cohort).

ELIGIBILITY:
Inclusion Criteria:

* indication for coronary CTA confirmed by board-certified radiologist ('justified indication' according to German/European radiation protection law) AND
* patient (is able to give informed consent and) has given informed consent.

Exclusion Criteria:

* contraindications to (iodine based) iv contrast material: known allergy to iodine-based iv contrast, acute or high-grade chronic kidney insufficiency with an estimated glomerular filtration rate < 30 ml/min/1.73 m², latent or manifest hyperthyroidism
* known or suspected pregnancy
* lactating mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are at least 18 years of age with a clincially indication for a coronary CTA scan. Indication ('justified indication' according to German/European radiation protection law) must be confirmed by a board-certified radiologist.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Intraluminal Enhancement of Coronary Arteries | 1 year
  measured on thin-slice reconstructions, in Hounsfield units
Image Noise | 1 year
  measured on thin-slice reconstructions, in Hounsfield units
Overall subjective image quality | 1 year
  as assessed by board-certified and speciality-trained radiologists on a 5-point Likert scale
Dose-Length Product (DLP) | 1 year
  Integrative descriptor for the x-ray dose applied during acquisition; can be read out from the scan protocol.

SECONDARY OUTCOMES:
Diagnostic Accuracy of Coronary Artery Stenosis Assessment in Comparison with invasive catheter angiography | 1 year
  Comparison in the subgroups of patients who als undergo invasive catheter angiography

CONTACTS AND LOCATIONS:
Overall Officials: Florian Schwarz, MD, Principal Investigator — University Hospital Augsburg

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data upon request (pending final approval by the data protection officer of the university hospital).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Requests for sharing individual participant data will be considered at the time of publication of the first manuscript containing result data.
Access Criteria: We plan to share data on request at this point in time.